CLINICAL TRIAL: NCT06361056
Title: A User-centered Mobile Health App to Promote Participation of Black Women in Breast Cancer Clinical Trials - Clinical Trial mHealth Study
Brief Title: Mobile Health App to Promote Participation of Black Women in Breast Cancer Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2140
Record Dates: First submitted 2024-03-22; First posted 2024-04-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: application; mHealth
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mHealth app (Experimental): Women enrolled in the mHealth app study will receive access to the "mHealth" app, a list of available clinical trials within a 50-mile radius of their zip code, and the existing standard of care packet of cancer center resources.
  Interventions: Behavioral: Survey; Behavioral: mHealth app

INTERVENTIONS:
Behavioral: Survey — All participants will complete a brief questionnaire.
  Other Names: Questionnaire
Behavioral: mHealth app — Eighty Black women with newly diagnosed breast cancer (inclusive of all stages) and who have access to a mobile device or computer will be recruited to the study intervention.

SUMMARY:
This study explores the overall feasibility, impact, and satisfaction of using the "mHealth app" on clinic workflow for Black or African American women diagnosed with breast cancer.

The "mHealth app" which can be used as a platform to share clinical trial education and communication, was created and tested in previous steps of this study.

DETAILED DESCRIPTION:
A patient advisory council (PAC) was recruited from established hospital and community networks (North Carolina Cancer Hospital's Patient and Family Advisory Board, and the Lineberger Community Outreach and Engagement Office's Community Advisory Board). The PAC informed the content of interview guides, questionnaire/survey instruments, and mHealth app design, and will be involved in the analyses of qualitative and quantitative data, and dissemination of study results.

After analysis of the in-depth interviews, the Connected Health for Applications and Interventions (CHAI) core staff developed a progressive web application "mHealth app". mHealth app was tested in a pilot study included 20 African American (AA) patients diagnosed with breast cancer were interviewed to answer questions that will better inform the clinical trial education and communication needs of Black women with breast cancer.

Eighty African American women with newly diagnosed breast cancer who have access to a mobile device or computer will be recruited for the study intervention. Women will receive access to the "mHealth" app, a list of available clinical trials within a 50-mile radius of their zip code, and the existing standard of care packet of cancer center resources. Participants will complete a brief questionnaire that will assess clinical trial knowledge, how often a clinical trial discussion occurred during their oncology appointment, and if a therapeutic trial was offered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Able and willing to participate to complete the survey.
* Have access to a mobile device or computer.
* Diagnosed with breast cancer.
* Identify as African American

Exclusion Criteria:

* Inability to read and speak English.
* Dementia altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are women with breast cancer
Enrollment: 80 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of Mobile Health Application (mHealth app)- subjects | Up to 1 year
  The feasibility of the mHealth app will be determined by the percentage of subjects who enrolled and completed trial requirements.
Feasibility of Mobile Health Application (mHealth app) - Clinicians and staff | Up to 1 year
  Clinicians and staff will be interviewed to assess feasibility.

SECONDARY OUTCOMES:
Overall satisfaction | Up to 1 year
  Overall satisfaction will be assessed by survey questions administered to study participants. The rate of participants' satisfactions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Marjory Charlot, MD, MPH, MSc, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials